CLINICAL TRIAL: NCT01401725
Title: Electronic Strategies to Enhance Venous Thromboprophylaxis in Hospitalized Medical Patients
Brief Title: Electronic Strategies to Enhance Venous Thromboemboli (VTE) Prophylaxis in Hospitalized Medical Patients
Acronym: E-SENTRY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Menaka Pai, Assistant Professor, McMaster University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HHS150411
Record Dates: First submitted 2011-07-19; First posted 2011-07-25 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Venous Thromboembolism
Keywords: venous thromboembolism; thromboprophylaxis; anticoagulants; hospitalized medical patients; electronic order sets; decision support; knowledge translation; patient safety
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Hamilton General Hospital (Experimental)
  Interventions: Behavioral: Electronic Order Entry System + CDSS
- Juravinski Hospital (Active Comparator)
  Interventions: Behavioral: Electronic Order Entry System Only
- St. Joseph's Hospital (Other)
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Electronic Order Entry System + CDSS — Physicians at this hospital will use an Electronic Order Entry System plus a computerized decision support system (CDSS) to support VTE prophylaxis decisions.
  Arms: Hamilton General Hospital
Behavioral: Electronic Order Entry System Only — Physicians at this hospital will use an Electronic Order Entry System
  Arms: Juravinski Hospital
Other: Usual Care — Physicians at this hospital will practice usual care (no Electronic Order Entry System and no CDSS for VTE prophylaxis decisions)
  Arms: St. Joseph's Hospital

SUMMARY:
Venous thromboemboli (VTE) are abnormal blood clots that commonly form in the blood vessels of the legs or lungs. They can block normal blood flow, damage organs, and even cause death. The risk of VTE is increased in people who are sick or immobile. VTE is the most common preventable cause of death in hospitalized patients, and its VTE prevention should be a top patient safety priority. Though there is good evidence that injectable blood thinners and/or compression stockings can prevent VTE, over 30% of hospitalized medical patients in Hamilton, Ontario receive inappropriate prevention. Hamilton Health Sciences Corporation is in the process of introducing "electronic order sets" - computer programs that help doctors order medications and other healthcare interventions for their patients. The investigators would like to study if these electronic order sets can help improve the rate of appropriate VTE prevention in hospitalized medical patients. The investigators will examine the rate before and after the introduction of electronic order sets at the Juravinski Hospital and the Hamilton General Hospital. Doctors at the Hamilton General Hospital will also get to use an additional computer program, called a computerized decision support system (CDSS), that helps them decide on the best strategy to prevent VTE in individual patients. The rates of VTE prevention at each hospital will be compared to each other, and to the rates at St. Joseph's Healthcare Hamilton, which will receive neither the order sets nor the CDSS.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients at least 18 years of age
* Hospitalization on a general internal medicine ward

Exclusion Criteria:

* Receiving therapeutic anticoagulation at time of hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2011-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Proportion of hospitalized medical patients who are appropriately managed for VTE prophylaxis | Participants will be followed for the duration of their hospital stay on a medical ward, an expected average of 5 days
  'Appropriate management' is defined as: (i) appropriate non-receipt of any form of prophylaxis when the patient has no VTE risk factors; (ii) appropriate receipt of pharmacologic prophylaxis when VTE risk factors are present and the patient has no contraindications for pharmacologic prophylaxis; or (iii) appropriate receipt of mechanical prophylaxis, when VTE risk factors are present and the patient has contraindications for pharmacologic prophylaxis.

SECONDARY OUTCOMES:
Hospital-acquired venous thromboembolism | Participants will be followed for 30 days, from the date of hospital admission
  VTE is defined as the presence of DVT or PE objectively confirmed by at least one of compression ultrasonography, venography, ventilation-perfusion lung scanning, CT pulmonary angiography, or a conventional pulmonary arteriogram.
  'Hospital-acquired' VTE is that which is not clinically evident or suspected at the time of admission, but is diagnosed during or up to 30 days after hospital admission.
Major bleeding | Participants will be followed for 30 days, from the date of hospital admission
  Major bleeding is defined using the International Society of Haemostasis and Thrombosis criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Menaka Pai, MD, FRCPC, Principal Investigator — McMaster University, Hamilton Health Sciences, Corporation - Hamilton General Hospital; James D Douketis, MD, FRCPC, Principal Investigator — McMaster University
Locations (3):
- Canada (3):
  - Hamilton General Hospital, Hamilton, Ontario
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Juravinski Hospital, Hamilton, Ontario

REFERENCES:
- [Background] Geerts WH, Bergqvist D, Pineo GF, Heit JA, Samama CM, Lassen MR, Colwell CW. Prevention of venous thromboembolism: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines (8th Edition). Chest. 2008 Jun;133(6 Suppl):381S-453S. doi: 10.1378/chest.08-0656. PMID 18574271
- [Background] Dentali F, Douketis JD, Gianni M, Lim W, Crowther MA. Meta-analysis: anticoagulant prophylaxis to prevent symptomatic venous thromboembolism in hospitalized medical patients. Ann Intern Med. 2007 Feb 20;146(4):278-88. doi: 10.7326/0003-4819-146-4-200702200-00007. PMID 17310052
- [Background] Kucher N, Koo S, Quiroz R, Cooper JM, Paterno MD, Soukonnikov B, Goldhaber SZ. Electronic alerts to prevent venous thromboembolism among hospitalized patients. N Engl J Med. 2005 Mar 10;352(10):969-77. doi: 10.1056/NEJMoa041533. PMID 15758007
- [Background] Durieux P, Nizard R, Ravaud P, Mounier N, Lepage E. A clinical decision support system for prevention of venous thromboembolism: effect on physician behavior. JAMA. 2000 Jun 7;283(21):2816-21. doi: 10.1001/jama.283.21.2816. PMID 10838650
- [Background] Garg AX, Adhikari NK, McDonald H, Rosas-Arellano MP, Devereaux PJ, Beyene J, Sam J, Haynes RB. Effects of computerized clinical decision support systems on practitioner performance and patient outcomes: a systematic review. JAMA. 2005 Mar 9;293(10):1223-38. doi: 10.1001/jama.293.10.1223. PMID 15755945